CLINICAL TRIAL: NCT01815671
Title: The Effect of Body Positioning for Colonoscopy in Women: Randomized, Study of Left Lateral Tilt Down Versus Left Lateral Horizontal Positioning
Brief Title: Evaluate the Safety and Diagnostic Advantages of Tilt Down Verses Standard Horizontal Colonoscopy Positioning
Acronym: CTDTTIE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Increased number of oxygen desaturation in tilt down position
Sponsor: Specialists in Gastroenterology, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: BP-1; Leonard Weinstock, MD (Other: Specialists in Gastroenterology)
Record Dates: First submitted 2013-03-18; First posted 2013-03-21 (Estimated); Results first posted 2014-02-05 (Estimated); Last update posted 2014-02-05 (Estimated); Status verified 2014-02

CONDITIONS: Diverticulosis
Keywords: colonoscopy; technique; tilt; insertion; safety; efficacy
MeSH Terms: conditions — Diverticulum | interventions — Colonoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lateral horizontal body position (Other): Subjects randomized to receive colonoscopy in the lateral horizontal position, This is the standard position. The other position - tilt down is the intervention
  Interventions: Procedure: colonoscopy in the lateral horizontal position
- Lateral tilt down body position (Other): Subjects randomized to receive colonoscopy in the lateral tilt down position
  Interventions: Procedure: colonoscopy in the lateral horizontal position

INTERVENTIONS:
Procedure: colonoscopy in the lateral horizontal position — colonoscopy in the lateral horizontal position with tilt down

SUMMARY:
A tortuous sigmoid colon makes colonoscopy difficult. The purpose of this study was to systematically evaluate the diagnostic utility and incidence of adverse events in women using standard horizontal compared to lateral tilt down positioning for colonoscopy.

DETAILED DESCRIPTION:
This was a prospective, randomized study. Subjects who provide informed consent and present to the offices of Specialists in Gastroenterology for colonoscopy will be randomized in a 1:1 distribution to either left lateral tilt down versus left lateral horizontal positioning to initiate colonoscopy.

Demographic data as well as routine information regarding the colonoscopy was filled out during or at the end of each procedure. In addition, the following parameters were assessed, and compared between groups:

1. Occurrence of complications related or possibly related to the colonoscopy procedure
2. Scope insertion time
3. Pain during and after the procedure

The subjects' participation was limited to the duration of the colonoscopy, which is typically less than 60 min and a follow up by telephone 24 hours later to assess the occurrence of complications.

ELIGIBILITY:
Inclusion Criteria:

* ability to understand and sign consent
* women and men with a BMI (body mass index) <35 kg/m2
* age 18 - 90 years
* no liquids by mouth for ≥2 hours
* no solid food for ≥8 hours

Exclusion Criteria:

* inability to provide informed consent
* morbid obesity (BMI ≥35)
* pregnancy
* uncontrolled gastroesophageal reflux disease
* gastroparesis
* scleroderma
* achalasia
* Crohn's disease
* ulcerative colitis
* history of a colon resection
* Parkinson's disease
* brain tumor
* multiple sclerosis
* ischemic optic neuropathy
* glaucoma
* active pulmonary infection
* liquid intake <2 hours
* solid food intake <8 hours prior to the procedure
* intra-procedure findings of a stricture resulting in an incomplete colonoscopy or Boston bowel preparation scores of <6

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2012-05; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonard B Weinstock, MD, Principal Investigator — Specialists in Gastroenterology, LLC
Locations (1):
- Advanced Endoscopy Center, St Louis, Missouri, United States

REFERENCES:
- [Background] Weinstock LB. Body positions for colonoscopy: value of Trendelenburg. Gastrointest Endosc. 2009 Jun;69(7):1409-10. doi: 10.1016/j.gie.2008.09.039. No abstract available. PMID 19481671

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Consecutive women presenting to a private endoscopy center for colonoscopy (with or without a preceding upper endoscopy) were offered participation. A computer generated randomization code was used to assign subjects to either TD or LL group. Subjects were blinded to which group they were assigned.
Pre-assignment Details: morbid obesity, pregnancy, uncontrolled gastroesophageal reflux disease, gastroparesis, scleroderma, achalasia, Crohn's disease, ulcerative colitis, history of a colon resection, Parkinson's disease, brain tumor, multiple sclerosis, ischemic optic neuropathy, glaucoma, active pulmonary infection
Groups:
- Lateral Horizontal: Subjects randomized to receive colonoscopy in the lateral horizontal position
- Lateral Tilt Down: Subjects randomized to receive colonoscopy in the lateral tilt down position
Period: Overall Study
Arm/Group | Lateral Horizontal | Lateral Tilt Down
Started | 88 | 85
Completed | 88 | 85
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lateral Horizontal | Lateral Tilt Down | Total
Number analyzed (Participants) | 88 | 85 | 173
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 4 | 7
  Between 18 and 65 years | 40 | 50 | 90
  >=65 years | 45 | 31 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (12) | 56 (11) | 55 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 85 | 173
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 88 | 85 | 173

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experience Adverse Events Which Are Related or Possibly Related to the Colonoscopy Procedure
Description: The number of participants who experience adverse events which are related or possibly related to the colonoscopy procedure will be tallied in each treatment arm.
Time Frame: 24 hours
Measure: Number; unit: participants
Arm/Group | Lateral Horizontal | Lateral Tilt Down
Number analyzed (Participants) | 88 | 85
participants | 2 | 9

2. Secondary Outcome: Time to Full Colonoscope Insertion
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Lateral Horizontal | Lateral Tilt Down
Number analyzed (Participants) | 88 | 85
minutes | 5.5 (1.2) | 5.2 (1.1)

3. Secondary Outcome: Pain Related or Possibly Related to Colonoscopy Procedure
Description: Visual Analogue Scale measured 0-4 with zero being no pain and 4 being most severe pain.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lateral Horizontal | Lateral Tilt Down
Number analyzed (Participants) | 88 | 85
units on a scale | 0.36 (0.03) | 0.28 (0.02)

ADVERSE EVENTS:
Arm/Group | Lateral Horizontal | Lateral Tilt Down
Serious Adverse Events (participants affected / at risk) | 0/88 | 0/85
Other Adverse Events (participants affected / at risk) | 2/88 | 9/85
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lateral Horizontal (N=88) | Lateral Tilt Down (N=85)
bradycardia (Cardiac disorders) | 2 (2) | 0 (0) — pulse less than 50 requiring medication
oxygen desaturation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 9 (9) — oxygen saturation less than 90 mm Hg for any length of time

LIMITATIONS AND CAVEATS:
Early termination owing to increased incidence of oxygen desaturation in the tilt down group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No